CLINICAL TRIAL: NCT05392374
Title: Expanded Access Use of ONC201 in a Patient With Diffuse Intrinsic Pontine Gliomas
Status: No longer available | Type: Expanded Access
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ONC016
Record Dates: First submitted 2021-12-01; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — TIC10 compound

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: ONC201 — ONC201 is an oral, small molecule selective antagonist of DRD2

SUMMARY:
This is an intermediate-size expanded access protocol to provide ONC201 to patients with diffuse intrinsic pontine gliomas who cannot access ONC201 through clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with DIPG who failed at least one line of prior therapy such as focal radiation therapy
2. Patient must be > than 6 months and < 18 years of age.
3. Confirmed evidence of disease progression from immediately prior therapy or refractory to the immediately prior treatment.
4. Karnofsky/Lansky performance status ≥ 50.
5. Adequate organ and marrow function as defined below:

   1. Absolute neutrophil count ≥1,000/mm3 without growth factor use ≤ 7 days prior to treatment (cycle 1 day 1, C1D1)

      ________________________________________________________________________________ CONFIDENTIAL Page 3 of 45
   2. Hemoglobin>8.0 mg/dL without red blood cell transfusion ≤ 3 days prior to C1D1
   3. Total serum bilirubin<1.5 X upper limit of normal (ULN)
   4. AST (SGOT)/ALT (SGPT)≤2 X ULN;; ≤ 5 X ULN if there is liver involvement secondary to tumor
   5. Serum creatinine≤ 1.5 X ULN (OR creatinine clearance ≥ 60 mL/min/1.73 m2)
6. Ability to understand and the willingness to sign a written informed consent document by the patient or their legal guardian.
7. If patient is of child--bearing age, female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. Male patients must be surgically sterile or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. The decision of effective contraception will be based on the judgment of the principal investigator or a designated associate.
8. Patient must be able to swallow capsules and retain orally administered medication.

Exclusion Criteria:

1. Body weight >10Kg.
2. Known active bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV).
3. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)--related illness.
4. Active or prior plasma cell leukemia (defined as either 20% of peripheral WBC comprised of plasma/CD138+ cells or an absolute count of 2 x 10^9/L).
5. Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia.
6. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism.
7. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or in the judgment of the investigator would make the patient inappropriate for entry into the study.

Ages: 6 Months to 18 Years
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - University of California San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - NYU Langone Health, New York, New York
  - Stephen Hassenfeld Children's Center for Cancer and Blood Disorders (NYU), New York, New York
  - University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Derived] Arrillaga-Romany I, Gardner SL, Odia Y, Aguilera D, Allen JE, Batchelor T, Butowski N, Chen C, Cloughesy T, Cluster A, de Groot J, Dixit KS, Graber JJ, Haggiagi AM, Harrison RA, Kheradpour A, Kilburn LB, Kurz SC, Lu G, MacDonald TJ, Mehta M, Melemed AS, Nghiemphu PL, Ramage SC, Shonka N, Sumrall A, Tarapore RS, Taylor L, Umemura Y, Wen PY. ONC201 (Dordaviprone) in Recurrent H3 K27M-Mutant Diffuse Midline Glioma. J Clin Oncol. 2024 May 1;42(13):1542-1552. doi: 10.1200/JCO.23.01134. Epub 2024 Feb 9. PMID 38335473